CLINICAL TRIAL: NCT05811091
Title: Prevalence of Pathological Patterns in Patients of Chronic Diarrhea With Normal Colonoscopy
Brief Title: Pathological Patterns in Chronic Diarrhea With Normal Colonoscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Mansour Omar, Clinical professor, Assiut University
Other Study IDs: Chronic diarrhea
Record Dates: First submitted 2023-03-16; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Chronic Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To asses prevalence of pathological findings in patients with chronic diarrhea and normal colonoscopy

DETAILED DESCRIPTION:
diarrhea is defined as the of 3 or more loose or liquid stools per day, or more frequently than is normal for the individual. 3. (World Health ion. Diarrhoeal disease .Available 2017) Diarrhea can be separated into acute, persistent and chronic types based on duration. Acute diarrhea lasts less than 14 days whereas persistent diarrhea is longer than 14 days, but no longer than 28 days( Zilla GC, Israel EJ. et al ..2012) Chronic diarrhea than 28 days. (Schiller LR, Parda DS, et al..2017) In addition to duration of symptoms, chronic diarrhea also tends to occur without a clear onset whereas persistent diarrhea can be thought of as an acute process that has persisted for a longer period.( zilla GC, Israel EJ. et al ..2012) it can be secondary to such heterogeneous causes as drug side effects, structural abnormalities of the small bowel and/or colon, the result of previous gastrointestinal surgery, inflammatory or neo-plastic pancreato biliary disease, or as part of an intestinal functional disorder, such as functional diarrhea, or irritable bowel syndrome (IBS) that is diarrhea predominant (IBS-D)or post infectious (PI-IBS) ( Burgers K, Lindberg B, 2020) or Primary eosinophilic colitis (PEC) is defined as an inflam-matory disease of unknown etiology that mainly manifests as abdominal pain and diarrhea, segmental or diffuse infil-tration of eosinophils in the mucosa of the colon,( Villanueva MS, Alimi Y.et al ..2015)( Impellizzeri G, Marasco G ,et al ..2019) or Enteropathies( are diseases that affect small bowel (SB) function and clinically manifest as chronic diarrhea).( Jansson-Knodell CL, Hujoel IA, et al 2017) as Monomorphic epitheliotropic intestinal T-cell lymphoma(MEITL) is a rare aggressive disease that mainly affects the SuB mucosa. Its symptoms can be nonspecific, but often presents chronic diarrhea (Ramírez-Quintero JD, Carvajal JJ,et al..2021) Evaluation of the colonic mucosa is very helpful in detecting inflam-matory bowel disease, ischemic colitis, microscopic colitis, neoplasis, and intraepithelial infections. The endoscopic appearance of the colon is normal, or almost normal, in some of those diseases, and thus they can go by un detected .Different studies have shown that systematic endoscopic biopsies of the colon provide good diagnostic yield in patients with chronic non inflammatory diarrhea and normal colonoscopy (López-Valenzuela LA, Murcio-Pérez E, et al..2019) chronic inflammatory disorder of the large intestine that mainly affects the elderly. Microscopic colitis differs from classical inflammatory bowel disease (IBD) in its almost normal-appearing colonic mucosa and histological findings consistent with increased lymphocytic infiltrates with or without collagen fiber expansion (Khalili et al., 2020). Microscopic colitis has two major subtypes, lymphocytic colitis (LC) and collagenous colitis (CC) (Shor et al., 2019) chronic watery diarrhea and often have no weight loss These forms of colitis also have an entirely of normal endoscopic appearance (Macaigne et al., 2014). If colonoscopy is done in patients suspected of having IBS-D, random colon biopsies should be done to rule out , structural abnormalities of the small bowel and/or colon, the result of previous gastrointestinal surgery, inflammatory or neo-plastic pancreato biliary disease, or as part of an intestinal functional disorder, such as functional diarrhea, or irritable bowel syndrome (IBS) that is diarrhea predominant (IBS-D)or post infectious (PI-IBS) ( Burgers K, Lindberg B, 2020) or Primary eosinophilic colitis and microscopic colitis (Münch et al., 2020).

ELIGIBILITY:
Inclusion Criteria:

* all patients with chronic diarrhea and had normal colonoscopy

Exclusion Criteria:

* Inflammatory bowel diseases (ulcerative colitis, crohns disease and indeterminate colitis).
* Systemic disease associated with chronic diarrhea, e.g. Diabetes mellitus and Thyroid disease.
* Drugs causing chronic diarrhea, e.g. antibiotics, antidepressants and angiotensin converting enzyme inhibitors.
* Chronic diarrhea due to decreased digestion as in pancreatic insufficiency,bile acid deficiency and Infectious colitis

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients from 18 to 75 years presented to out patient clinic in Elraghi hospital in Assuit university with chronic diarrhea and normal colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-05 (Estimated); Primary Completion 2024-03-06 (Estimated); Study Completion 2024-05-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of pathological patterns in patients of chronic diarrhea with normal colonoscopy | 1year
  As number of patients who has chronic diarrhea and thier colonoscopy was normal we need to know pathological pattern in thier biopsies if esinophilic or lymphcytic and either